CLINICAL TRIAL: NCT01432964
Title: Low Profile Titanium Mesh in the Use of Orbital Reconstruction
Brief Title: Use of a Low Profile Titanium Mesh in Orbital Reconstruction
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: International Bone Research Association (Other)
Responsible Party: Principal Investigator Olivier Lieger, Department of Oral and Maxillofacial Surgery, University Hospital Bern, Switzerland
Other Study IDs: 011/09; 0709-0050
Record Dates: First submitted 2011-09-12; First posted 2011-09-13 (Estimated); Last update posted 2011-09-13 (Estimated); Status verified 2011-09

CONDITIONS: Orbital Fractures
Keywords: Orbital Fractures; Fracture Fixation; Blow-out Fractures; Surgical Mesh; Titanium; Computer-assisted Image Processing
MeSH Terms: conditions — Orbital Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Adult patients (>18 years) presenting a unilateral orbital blow-out or blow-in fracture of ≥ 2.0cm2, causing an actual or expected functional or aesthetical deficit.
  Interventions: Procedure: Orbital revision surgery

INTERVENTIONS:
Procedure: Orbital revision surgery — Surgical revisions were performed under general anaesthesia. The orbital floor was routinely exposed via a transconjunctival incision. In patients with involvement of the medial wall, a combined transconjunctival-transcaruncular approach was used. Herniated or incarcerated tissue was then complete repositioned. Stable borders around the bony defect in the orbital floor were exposed. The aluminium template was pre-bend and controlled in situ. Type and size of mesh were chosen and adjustments performed, as needed. Following the bending of the titanium mesh according to the template, it was inserted and fixed with 1.5mm screws. Alternatively the mesh could be preformed, using a sterilized skull model to shape and contour it to a normal orbit. Finally the eye bulb mobility was controlled using fine forceps (forced duction test) and the wound closed (Vicryl 5/0 rapid; optional).

SUMMARY:
In craniofacial trauma, the involvement of orbital structures is noted in up to 40% of cases (Ellis 1985). Post-traumatic orbital deformities caused by incorrect reconstruction of orbital dimensions are severe complications causing enophthalmos, diplopia and visual acuity disturbance. To prevent such complications, immediate repair of orbital injuries with the restoration of normal anatomy is indicated in orbital floor fractures. With the help of biodegradable implants small and medium-sized defects are easily managed (Büchel 2005, Lieger 2010). In extensive fractures however, only calvarian bone and titanium mesh considered to provide a sufficient support of the orbital content.

Calvarial bone can be difficult to mould and to adapt to the form and size of the orbital lesion. In addition, donor site morbidity cannot be disregarded. Orbital reconstruction mesh on the other hand is always available and easier to apply. There are however important requirements for these meshes, such as biocompatibility, excellent stability, optimal adaptability and patient comfort. Recently, the company Medartis developed a titanium mesh featuring a low profile. In order to regain normal function, normal anatomy has to be re-established. It therefore seemed reasonable to assess an implant, which would facilitate orbital reconstruction without disturbing normal anatomy by its size, profile height or properties.

The purpose of this study was to assess the use and accuracy of the low profile titanium mesh for primary internal orbital reconstruction.

DETAILED DESCRIPTION:
Background

Extensive bone loss after orbital trauma requires reconstruction to preserve ocular function and aesthetics. The optimal material for orbital reconstruction remains controversial. Today a multitude of both autogenous and alloplastic materials have been used for orbital reconstruction, including methylmethacrylate, Teflon, silicone, Supramid, Marlex, Silastic, gelatin film, bioactive glas, bone and cartilage (Haug 1999). The use of alloplastic materials has been tempered by complications such as infection, displacement and extrusion, fistula and cyst formation. During the past two decades, autogenous bone grafts have become increasingly popular for orbital reconstruction. Unfortunately, problems with bone grafts can occur and include unpredictable rates of bone resorption and the risk of subsequent dystopia or delayed enophthalmos, donor site complication, time consumption with harvesting and variable graft thickness and irregularities along with difficulty in graft contouring (Park 2001). These problems have revived interest in alloplastic alternatives, particularly in titanium and its alloys (Park 2001). Titanium shows a low infection rate, related in part to its excellent biocompatibility, which manifests as osseointegration. This circumstance is thought to lessen the rate of infection.

During the past decade, different studies have examined a titanium meshes for orbital repair. Plates used in these studies demonstrate a minimum profile height of 0.25mm.

Objective

Assess the use and accuracy of the low profile titanium mesh for primary internal orbital reconstruction

Methods

Clinical assessment prior to operation by a maxillofacial surgeon with regards to bone and soft tissue lesions as well as concomitant injuries. An ophthalmologist then assessed eye lesions and quantified eye mobility (in mm), bulb positioning (Hertel's exophthalmometry, in mm) as well as the field of binocular vision (Goldmann perimetry, in % of the total).

Preoperative 1mm CT-scans were obtained to analyse size and location of the defect as well as extend of muscle entrapment. The fractures were classified according to the scores introduced by Jaquiery(Jaquiery 2007).

Follow up by at 2, 6 and 12 weeks after the operation (assessments see above), including postoperative CT-scan within 12 weeks. Volume analysis of CT comparing the two orbits (OsiriX Medical Image Software (Version 3.7.1, www.osirix-viewer.com).

ELIGIBILITY:
Inclusion Criteria:

* adult patients (>18 years)
* presenting a unilateral orbital blow-out or blow-in fracture of ≥ 2.0cm2, causing an actual or expected functional or aesthetical deficit
* has to be operated within two weeks of trauma

Exclusion Criteria

* individuals who did not have any vision on the affected side
* individuals, who, according to ophthalmologists, should not have a surgical treatment
* patients who were unable to adequately understand written or oral information in German or French

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with facial fractures, treated at the Department of Oral and Maxillofacial Surgery, University Hospital Bern, Bern, Switzerland.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2008-12; Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Radiological Volume analysis of bony orbits (difference in cm3) | postoperative, within 12 weeks after operation

SECONDARY OUTCOMES:
Eye motility (in mm) | at 12 weeks after the operation
En/Exophthalmos (Hertel Test) (in mm) | at 12 weeks after the operation
Diplopia (in %) | at 12 weeks after the operation

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Lieger, MD, DMD, Principal Investigator — Department of Oral and Maxillofacial Surgery, University Hospital Bern, Switzerland; Tateyuki Iizuka, MD, DDS, PhD, Study Director — Department of Oral and Maxillofacial Surgery, University Hospital Bern, Switzerland
Locations (1):
- Department of Oral and Maxillofacial Surgery, Bern University Hospital, Bern, Switzerland

REFERENCES:
- [Background] Ellis E 3rd, el-Attar A, Moos KF. An analysis of 2,067 cases of zygomatico-orbital fracture. J Oral Maxillofac Surg. 1985 Jun;43(6):417-28. doi: 10.1016/s0278-2391(85)80049-5. PMID 3858478
- [Background] Buchel P, Rahal A, Seto I, Iizuka T. Reconstruction of orbital floor fracture with polyglactin 910/polydioxanon patch (ethisorb): a retrospective study. J Oral Maxillofac Surg. 2005 May;63(5):646-50. doi: 10.1016/j.joms.2004.11.013. PMID 15883939
- [Background] Lieger O, Schaller B, Zix J, Kellner F, Iizuka T. Repair of orbital floor fractures using bioresorbable poly-L/DL-lactide plates. Arch Facial Plast Surg. 2010 Nov-Dec;12(6):399-404. doi: 10.1001/archfacial.2010.91. PMID 21079117
- [Background] Haug RH, Nuveen E, Bredbenner T. An evaluation of the support provided by common internal orbital reconstruction materials. J Oral Maxillofac Surg. 1999 May;57(5):564-70. doi: 10.1016/s0278-2391(99)90076-9. PMID 10319830
- [Background] Park HS, Kim YK, Yoon CH. Various applications of titanium mesh screen implant to orbital wall fractures. J Craniofac Surg. 2001 Nov;12(6):555-60. doi: 10.1097/00001665-200111000-00010. PMID 11711822
- [Background] Jaquiery C, Aeppli C, Cornelius P, Palmowsky A, Kunz C, Hammer B. Reconstruction of orbital wall defects: critical review of 72 patients. Int J Oral Maxillofac Surg. 2007 Mar;36(3):193-9. doi: 10.1016/j.ijom.2006.11.002. Epub 2007 Jan 22. PMID 17241771